CLINICAL TRIAL: NCT05057663
Title: Intralesional Injection of Bleomycin Versus 5-fluorouracil in Treatment of Plantar Wart; a Comparative Study
Brief Title: Intralesional Treatment of Plantar Wart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rania Farouk Daif, Director, Head of Dermatology, Andrology and Venerology, Principal investigator, clinical professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-09-03
Record Dates: First submitted 2021-09-12; First posted 2021-09-27 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Plantar Wart
Keywords: Intralesional Injection.; Bleomycin.; 5-Fluorouracil.
MeSH Terms: interventions — Bleomycin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bleomycin group (Active Comparator)
  Interventions: Drug: Bleomycin and 5-fluorouracil
- 5-Fluorouracil group (Active Comparator)
  Interventions: Drug: Bleomycin and 5-fluorouracil

INTERVENTIONS:
Drug: Bleomycin and 5-fluorouracil — In the bleomycin-treated group, bleomycin vial will be diluted first with 5 ml distilled water At time of treatment session 2 ml of lidocaine 2% and 1 ml of the bleomycin stock solution will be taken in 100-unite insulin syringe. Thus, the working bleomycin solution will be used in treatment 1 mg/ml. The bleomycin solution will be injected intralesional till blanching of the wart will be occurred. The amount of injection ranging from 0.2, 0.5, 1 ml according to size of warts; (5 mm, 10 mm, >10 mm) maximum for 1 ml in single wart and 2ml in treatment session. Treatment session will be done every two weeks maximum four sessions.
  In 5-fluorouracil treated group, 5-fluorouracil vial ( 1 ml of 50 mg/ml 5-FU will be mixed with 0.25 ml of lidcaine 2% Every wart will be injected with 0.1 ml of the previous mixture into it base using an insulin syringe till blanching of the warts maximum 2ml of 5-FU per session. Treatment session will be done every two week for maximum 6 sessions

SUMMARY:
Group 1; intralesional injection of bleomycin in plantar wart. Group 2; intralesional injection of 5-fluorouracil in plantar wart

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be considered for participation in this study.

1. Subject is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
2. Male or female ≥ 8 years old.
3. Subject has a clinical diagnosis of common warts.
4. Subject has up to 1 Target Wart and up to 3 additional Non-Target Warts located on the trunk or extremities. The identified Target and Non-Target Warts must meet the requirements as defined below:

   1. Each wart must have a longest axis that is ≥ 3mm and ≤ 8 mm and have a thickness of ≤3mm
   2. Each wart must be a discrete lesion
   3. Each wart must be present for at least 4 weeks
   4. Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   5. Not be in an intertriginous fold
   6. Be the only common wart present when the circular cutout template is centered over the wart
5. The Target and Non-Target Warts must have a PWA ≥ 2.
6. Subject chemistry and complete blood count results are within normal limits. If any of the laboratory values are outside normal range, the treating investigator must assess the value/s as NOT clinically significant and document this in the subject's medical chart in order for the subject to be eligible for randomization.
7. Woman of childbearing potential (WOCBP) must have a negative urine pregnancy test within 14 days of the first application of study drug and agree to use an active method of birth control for the duration of the study.
8. Subject is non-pregnant and non-lactating.
9. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of any Target or Non-Target Warts or which exposes the subject to an unacceptable risk by study participation.
10. Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

Subjects are excluded from this study if any 1 or more of the following criteria is met:

1. Subject has clinically atypical warts on the trunk or extremities.
2. Subject is immunocompromised (e.g., due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Response to intralesional injection of bleomycin, 5fluorouracil in treatment of plantar wart | 3monthes
  Physician's Wart Assessment Grade Descriptor 0 Clear: No visible wart. No further treatment is indicated
  1. Near Clear: A visible wart that is less than 3mm in maximal diameter (or length)
  2. A visible wart ≥ 3mm and <6 mm in maximal diameter (or length)
  3. A visible wart ≥ 6mm in maximal diameter (or length)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Farouk, Resident, Principal Investigator — Sohag Faculty of medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt